CLINICAL TRIAL: NCT02406274
Title: Use of Contrast Enhanced Spectral Mammography (CESM) for Women With Palpable Breast Abnormalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-053
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Breast Abnormalities
Keywords: Mammography; Contrast Enhanced Spectral Mammography; Palpable Breast Abnormalities; 15-053

ARMS (1):
- Contrast Enhanced Spectral Mammography (Experimental)
  Interventions: Other: Contrast Enhanced Spectral Mammography (CESM)

INTERVENTIONS:
Other: Contrast Enhanced Spectral Mammography (CESM) — Women presenting to MSKCC with a palpable abnormality within the breast either self palpated & or palpated by their physician will be offered CESM instead of FFDM alone. The breast imager assigned to care for the patient will interpret the low energy images (including any additional views they routinely obtain) & record their findings. They will then interpret the CESM & record those results. As per standard of care, the patient will have a targeted ultrasound as well. Appropriate clinical recommendations will be made. In patients with no specific imaging findings, follow-up will be determined by the degree of suspicion of the palpable finding & will either be called negative & followed clinically if not suspicious, or will go on to MRI , percutaneous biopsy by a surgeon or surgical biopsy if suspicious.

SUMMARY:
Contrast Enhanced Spectral Mammography (CESM) is an advanced form of mammography which is performed after injection of contrast or dye into a vein in the arm. This dye is the same dye that is used for CT scans. This type of mammogram includes a regular mammogram as well as additional pictures with the dye.

This particular study is being done to determine if by adding the dye in the veins the investigators are better able to identify the cause of the lump than if they just did the regular mammogram alone.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting for mammographic evaluation of an undiagnosed palpable mass found either by self examination and/or examination by referring physician

Exclusion Criteria:

* Age < 25 years old
* Male patients
* Pregnant or lactating patients
* Patients with allergy to iodinated contrast
* Patients with a history of renal disease or patients over 70 with a creatinine > 1.3. Creatinine must have been done within the last 12 weeks.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
positive predictive value | 1 year
  (PPV) will be defined using three distinct definitions: (1) PPV1 is the proportion of women with a positive assessment who had a cancer diagnosis in the follow-up period. (2) PPV2 is the proportion of women with a recommendation for biopsy who had a cancer diagnosis in the follow-up period. (3) PPV3 is the proportion of women with a biopsy recommendation and a biopsy performed within 1 year who had a cancer diagnosis in the follow-up period. Negative predictive value (NPV) is the proportion of women with a negative assessment who did not have a cancer diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Maxine Jochelson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/